CLINICAL TRIAL: NCT03035318
Title: Comparison of Glenoid Position Using SmartBones: A Randomized Clinical Trial
Brief Title: Comparison of Glenoid Position Using SmartBones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joseph Iannotti, Chairman, Orthopaedic and Rheumatologic Institute, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-789
Record Dates: First submitted 2017-01-18; First posted 2017-01-30 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: Anatomic Total Shoulder Arthroplasty
Keywords: Anatomic Total Shoulder Arthroplasty; Glenoid; Patient-specific instrumentation; Computer simulation; Computer assisted tomography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- DePuy Global® Anchor Peg Glenoid (Active Comparator): In the setting of Anatomic Total Shoulder Arthroplasty, this arm uses DePuy Global® Anchor Peg Glenoid Instrumentation to position the glenoid component.
  Interventions: Device: DePuy Global® Anchor Peg Glenoid Instrumentation
- DePuy Instrumentation with SmartBone™ (Experimental): In the setting of Anatomic Total Shoulder Arthroplasty, this arm uses DePuy Global® Anchor Peg Instrumentation with SmartBone™, to position the glenoid component.
  Interventions: Device: DePuy Global® Anchor Peg Instrumentation with SmartBone™
- IRI with SmartBone™ (Experimental): In the setting of Anatomic Total Shoulder Arthroplasty, this arm uses an Intelligent Reusable Instrumentation (IRI), with a SmartBone™, to position the glenoid component.
  Interventions: Device: IRI with SmartBone™
- RTI with SmartBone™ (Experimental): In the setting of Anatomic Total Shoulder Arthroplasty, this arm uses Real Time Instrumentation (RTI), with a SmartBone™, to position the glenoid component.
  Interventions: Device: RTI with SmartBone™
- IRI with SmartBase (Experimental): In the setting of Anatomic Total Shoulder Arthroplasty, this arm uses an Intelligent Reusable Instrumentation (IRI), with a SmartBase™, to position the glenoid component.
  Interventions: Device: IRI with SmartBase

INTERVENTIONS:
Device: DePuy Global® Anchor Peg Glenoid Instrumentation — Placement of glenoid component will be performed using DePuy Global® Anchor Peg Glenoid Instrumentation.
  Arms: DePuy Global® Anchor Peg Glenoid
Device: DePuy Global® Anchor Peg Instrumentation with SmartBone™ — Placement of glenoid component will be performed using DePuy Global® Anchor Peg Instrumentation with SmartBone™.
  Arms: DePuy Instrumentation with SmartBone™
Device: IRI with SmartBone™ — Placement of glenoid component will be performed using Intelligent Reusable Instrumentation (IRI) with SmartBone™.
  Arms: IRI with SmartBone™
Device: RTI with SmartBone™ — Placement of glenoid component will be performed using Real Time Instrumentation (RTI) with SmartBone™.
  Arms: RTI with SmartBone™
Device: IRI with SmartBase — Placement of glenoid component will be performed using Intelligent Reusable Instrumentation (IRI) with SmartBase.
  Arms: IRI with SmartBase

SUMMARY:
The investigators propose a randomized clinical trial to evaluate the accuracy of glenoid implant placement comparing four groups of patients. Group 1 consists of 3D imaging and computer-generated surgical planning using standard DePuy instrumentation for placement of the glenoid implant. This group is considered the standard of care. Group 2 consists of 3D imaging and computer-generated surgical planning, with use of a SmartBone to trial the standard DePuy instrumentation. (Group 2 is Group 1 with addition of the use of a SmartBone.) Group 3 consists of 3D imaging and computer-generated surgical planning, with use of the IRI technology including a SmartBone, but with metal legs instead of plastic legs in the IRB#13-652 study. Group 4 consists of 3D imaging and computer-generated surgical planning, with use of the RTI technology including a SmartBone.

We will measure implant placement based on 3D CT imaging. We will measure pre-operative bone quality using quantitative CT scan to measure trabecular bone volume and correlate these findings with bone samples removed from the humeral head and measured by microCT and mechanical testing of the bone samples. These bone samples will be obtained as part of the routine preparation of the humeral head for implant placement. This bone tissue is normally removed and discarded as part of the standard of care for preparation of the bone for placement of the humeral stem.

By comparing a computer generated pre-operative plan to the post-operative glenoid component placement, we will be looking at three outcomes. First, we will determine the overall difference in glenoid component placement between the four treatment groups. Second, we will compare the placement between the technologies within and among surgeons. Third, we will evaluate the difference in implant position between technologies based on severity of pathology. The quality of the humeral head sample will be correlated to the possible loosening of the implants.

DETAILED DESCRIPTION:
The proposed clinical study will enroll patients indicated for standard of care anatomic total shoulder arthroplasty. Participants will receive all pre-operative testing, intra-operative care including all implants and post-operative care that is standard of care and specific to the surgeon's and patient's decisions for care. The only change for Groups 2, 3 and 4 will be the type of surgical instruments used to place the glenoid guide pin, retention of the humeral head to obtain bone tissue, placement of the beads and post-operative CT scanning. In all cases the surgeon is able and allowed to use their own surgical judgment to place the guide pin, prepare the bone and place the desired implant. In all cases, the surgeon can use any and all of the standard instruments or guides provided by the implant manufacturer as the surgeon would use if the patient was not enrolled in the study. If the surgeon chooses not to use the IRI or RTI technology, then this would be noted as a deviation in plan, the reasons recorded and the patient would be excluded from the study without post-operative imaging and their pre-operative and intra-operative data would be analyzed for the purpose of understanding the reasons for failure of the IRI or RTI technology to provide assistance for refinement of the technology.

The participating surgeons will be Dr. Joseph Iannotti, Dr. Eric Ricchetti and Dr. Peter Evans. Patients may have surgery at either Cleveland Clinic main campus or at Euclid Hospital. If the procedure is performed at Euclid Hospital, post-operative CT scan and RSA (if chosen), will be performed at main campus within 3 weeks after surgery. The patient will be made aware of this at the time of enrollment and consent.

Using manufacturer (RSA biomedical, Umsa Sweden) provided beads and injector gun, four to five 1 mm tantalum beads will be placed in the coracoid, acromion and glenoid. Exact placement of these beads is at the discretion of the surgeon. Patient anatomy and operative exposure will guide the surgeon to the best places to inject the beads; however the surgeon will not be confined to a specific amount of beads in a specific location. The beads just need to be spread out amongst the coracoid, acromion, and glenoid to establish reference points for the RSA imaging. Prior studies looking at shoulder joint kinematics and implant position have used this methodology of bead placement with successful study related outcomes. Investigators have successfully placed bone beads in 22 patients currently treated in the ongoing IRI clinical study without any difficulty or adverse events during or after surgery.

Postoperatively, all patients will receive a CT with Metal Artifact Reduction (MAR)and RSA (if chosen) within 3 weeks of surgery. This will be a CT Scan performed with the patient's arm by the side in a supine position using metal artifact reduction techniques. In addition patients will receive a second CT scan and RSA imaging, provided they originally got RSA, performed 1 year (± 1 month) from surgery. The second CT scan will be performed with MAR techniques and with the patient in the lateral decubitus position with their arm in the overhead position, again using metal artifact reduction techniques. The second set of images, produced with a different body and arm position, also decreases metal artifact than those obtained with the arm placed by the side. This position cannot be comfortably obtained until 3- 6 months after surgery and require healing of the tissues and rehabilitation of the shoulder. Investigators have shown that in a small number of patients the glenoid component can shift in position within the first 3-6 months after surgery making the first CT Scan more accurate for implant position. The images obtained from the postoperative CT scans are placed back into the surgical software and the 3D reconstruction of the postoperative scapula with the implants is compared to the preoperative plan. Using measurement tools within the software, developed at the Cleveland Clinic, investigators will compare the position of the actual glenoid component placed in the patient with the desired position specified by the plan. The use and validation of these imaging methods to precisely measure implant position has been performed at the Cleveland Clinic in a prior IRB approved clinical trial (IRB 10-582).

Preoperatively, the high resolution quantitative CT will measure volumetric bone mineral density and the trabecular network of the glenoid. When available, this will be applied to the preoperative CT for those patients at Cleveland Clinic, Main Campus. Patients who have their preoperative CT completed at non Main Campus facilities will have the standard of care preoperative CT. This will be done at the same visit for the standard of care preoperative CT. Micro CT imaging, which creates a 3D reconstruction of the fine bone structure, in addition to microarchitecture analysis and mechanical testing, will allow assessment of the bone tissue taken from the bone core sample. Between the preoperative imaging and the bone tissue analysis, investigators will have data to properly determine the quality of the bone stock surrounding the implant. Further correlating these data with RSA and 3D CT imaging of implant movement, investigators can fully develop cause and effect of bone quality on glenoid component loosening.

Study Statistics and Analysis:

Our goal is to have 20 subjects in each of the 4 treatment groups for a total of 80 subjects. To control for subject withdrawal for various reasons after enrollment, we will enroll up to 120 subjects.

Statistical analysis plan:

Average deviations from plan for the 4 treatment groups will be compared using mixed-effects ANOVA methods. Random effects will be included to account for correlation between observations introduced as a consequence of multiple observations of deviation being taken on a particular surgeon. If significant differences are found, multiple comparisons based on the ANOVA model will be made to compare each pair of groups, and will use Holm's step-down procedure to control the family-wise error rate of the tests.

All analyses will be done by Colin O'Rourke of Quantitative Health Sciences at Cleveland Clinic using R software (version 3.0.0, Vienna, Austria). A significance level of 5% will be used for all testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glenohumeral osteoarthritis
* Anatomic Total Shoulder Arthroplasty

Exclusion Criteria:

* Age < 18 or > 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Iannotti, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase
Started | 24 | 25 | 25 | 25 | 27
Completed | 22 | 21 | 21 | 23 | 20
Not Completed | 2 | 4 | 4 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase | Total
Number analyzed (Participants) | 22 | 21 | 23 | 21 | 20 | 107
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 22 | 21 | 23 | 21 | 20 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 4 | 6 | 12 | 31
  Male | 15 | 19 | 19 | 15 | 8 | 76

OUTCOME MEASURES:

1. Primary Outcome: Difference in Glenoid Component Position (Inclination and Version)
Description: The overall distance between glenoid component placement between Standard Manufacturer Instrumentation and Patient Specific Instrumentation will be compared (Inclination and Version).
Time Frame: Four months post surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase
Number analyzed (Participants) | 22 | 21 | 23 | 21 | 20
degrees
  Inclination | 3.5 (3.0) | 3.0 (3.2) | 3.0 (2.6) | 2.5 (1.8) | 2.5 (1.8)
  Version | 3.9 (3.4) | 4.5 (3.9) | 4.0 (2.5) | 4.3 (3.3) | 3.7 (2.7)

2. Secondary Outcome: Accuracy of Glenoid Component Placement Based on Severity of Glenoid Morphology
Description: Accuracy of glenoid component placement based on severity of glenoid morphology. Each shoulder was classified according to a modified Walch classification. The Walch classification of glenoid morphology is the most commonly used system describing glenohumeral pathology in primary osteoarthritis. Glenoids were classified as asymmetric moderate-to severe posterior glenoid bone loss (Walch type-C or moderate to-severe type-B2 and B3 glenoids), without bone loss (Walch type-A1 glenoid), posterior bone loss requiring <10 degrees of correction (Walch type-B1 or mild type-B2 and B3 glenoids), or symmetric glenoid bone loss (Walch type-A2 glenoid).
Time Frame: Four months post surgery
Population: Outcome measures data not collected/ no patients analyzed for this OM.
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Difference in Glenoid Component Position (AP and IP)
Description: The overall distance between glenoid component placement between Standard Manufacturer Instrumentation and Patient Specific Instrumentation will be compared (Anteroposterior Position and Superoinferior Position).
Time Frame: Four months post surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase
Number analyzed (Participants) | 22 | 21 | 23 | 21 | 20
mm
  Anteroposterior Position | 1.2 (0.8) | 1.5 (0.9) | 1.1 (0.8) | 1.5 (1.1) | 1.1 (0.9)
  Superoinferior Position | 1.2 (1.1) | 1.4 (0.9) | 1.6 (1.0) | 1.3 (0.9) | 1.1 (0.9)

ADVERSE EVENTS:
Time Frame: Approximately 1 year from the time of surgery.
Description: Adverse events include excessive bleeding, infection, fracture nerve injury or need for revision surgery during the term of this study which is expected to be approximately 1 year from the time of surgery. All-cause mortality was not monitored/assessed for this study.
Arm/Group | DePuy Global® Anchor Peg Glenoid | DePuy Instrumentation With SmartBone™ | IRI With SmartBone™ | RTI With SmartBone™ | IRI With SmartBase
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/23 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/23 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT03035318/Prot_SAP_000.pdf